CLINICAL TRIAL: NCT04314739
Title: The Acute and Chronic Effects of Resveratrol Supplementation on Inflammation and Cognitive Performance in Healthy Adults
Brief Title: The Effects of Resveratrol Supplementation on Inflammation and Cognitive Performance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Evolva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 52P7
Record Dates: First submitted 2019-04-01; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Change; Mood; Systemic Inflammation
Keywords: Resveratrol; Polyphenol; Cognition; Mood; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Active Comparator): 500mg of Veri-te Resveratrol (consumed as two 250mg tablets, at two timepoints each day).
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Matched placebo capsules (1 capsule consumed at two timepoints each day).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Participants will consume one of the treatment types daily for a period of four weeks.
  Other Names: Veri-teTM Resveratrol
  Arms: Resveratrol
Dietary Supplement: Placebo — Participants will consume one of the treatment types daily for a period of four weeks.
  Arms: Placebo

SUMMARY:
Previous research has suggested that high levels of systemic inflammation can contribute to cognitive deficits and additional health problems; consumption of polyphenols have been shown to have an anti-inflammatory effect. Resveratrol, a polyphenol found primarily in red grape skins, has previously been shown to improve brain blood flow and possibly brain function and may potentially reduce systemic inflammation, however there is limited research into this.

This study will investigate the effects of 4 weeks daily consumption of resveratrol on inflammation and cognitive function in healthy adults.

DETAILED DESCRIPTION:
Each participant will be required to attend the laboratory on three occasions. The first of these will be an initial screening/training visit, this will take place in the afternoon and last 2 1/2 hours in total. During the initial visit participants will be asked to provide written informed consent. They will provide lifestyle and demographic data and screened regards to physical health (height, weight, blood pressure, waist to hip ratio). They will then complete a food frequency questionnaire and be trained on the computerised cognitive and mood tasks. Participants will also be trained on completing the cognitive assessment battery on their mobile phone, they will complete a further 5 assessments on their phone, once the day before their first visit and every 7 days during the supplementation period.

Study days 1 and 2 (4 weeks apart) :

Participants will arrive at the laboratory at an agreed time in the morning (7am, 8.30am or 10am) having fasted for 12 hours, avoided caffeinated products for 18 hours, alcohol and over the counter medication for 24 hours and oral antihistamines for 48 hours prior to the session commencing.

Participants will provide a blood sample, they will then complete a short computerised cognitive assessment (~20 minutes in length), followed by measurements of blood pressure and heart rate. Following this the participants will consume their treatment for the day, followed by a 40 minute absorption period and then will complete the second cognitive assessment. Participants will then provide a second blood sample. At the end of the first study session participants will be provided with their treatment and treatment diary, they will be instructed to take one tablet twice a day (30 minutes after breakfast and dinner). Both study visits will be identical and will take place 29 days (+/- 2 days) apart.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health.
* Aged 18 to 55 at the time of giving consent

Exclusion Criteria:

* Have a Body Mass Index (BMI) outside the range of 18.5-42kg/m2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline concentration of biomarkers of systemic inflammation | 1 hour post dose; 4 weeks
  Assessment of change from baseline: C reactive protein, tumor necrosis factor alpha and interleukin 6.

SECONDARY OUTCOMES:
Acute changes in cognitive task performance | 40 minutes post dose
  This will be assessed using a computerised cognitive battery (administered using COMPASS cognitive assessment program). Changes in episodic memory, working memory, spatial memory, executive function and attention as compared to pre-treatment performance on day 1. All tasks have the same x3 outcome measures; accuracy (% correct), errors (% incorrect) and speed (milliseconds) and the individual task scores will therefore be collapsed into global cognitive domains.
Interim changes in cognitive task performance | Day 7; Day 14; Day 21; Day 28
  This will be assessed using a computerised cognitive battery, this will be administered using 'Cognimapp'mobile phone program, participants will complete this battery away from home using their own mobile phone. Changes in attention, executive function, working memory and episodic memory as compared to performance on Day -1. All tasks have the same x3 outcome measures; accuracy (% correct), errors (% incorrect) and speed (milliseconds) and the individual task scores will therefore be collapsed into global cognitive domains.
Chronic changes in cognitive task performance | 4 weeks
  This will be assessed using a computerised cognitive battery (administered using COMPASS cognitive assessment program). Changes in episodic memory, working memory, spatial memory, executive function and attention as compared to pre-treatment performance on day 1. All tasks have the same x3 outcome measures; accuracy (% correct), errors (% incorrect) and speed (milliseconds) and the individual task scores will therefore be collapsed into global cognitive domains.
Acute changes in mood | 40 mins post dose
  Assessed using Visual Analogue Mood Scales at each assessment during each cognitive assessment. Participants will complete 27 separate visual analogue mood scales that load onto 3 mood outcomes: Alertness, Stress and Tranquillity (the individual scale results are averaged to create this score). A score between 0 and 100 can be obtained, where a higher value indicates that the participant felt more Alert, Stressed or Tranquil.
Interim changes in mood | Day 7; Day 14; Day 21; Day 28
  Assessed using Visual Analogue Mood Scales at each assessment during the interim supplementation period. Participants will complete 27 separate visual analogue mood scales that load onto 3 mood outcomes: Alertness, Stress and Tranquillity (the individual scale results are averaged to create this score). A score between 0 and 100 can be obtained, where a higher value indicates that the participant felt more Alert, Stressed or Tranquil.
Chronic changes in mood | 4 weeks
  Assessed using the Profile of Mood States questionnaire, completed at the start of each testing visit. The questionnaire includes 65 items and participants rate their mood on a scale of 0-4 (not at all - extremely). These scores are collapsed into 6 mood outcomes (Tension, depression, anger, vigour, fatigue and confusion) and a total mood disturbance score.
Acute changes in concentration of plasma and serum biomarkers | 1 hour post dose
  Biomarkers of insulin, glucose, cholesterol and resveratrol metabolites will be measured in plasma and serum using liquid chromatography-mass spectrometry and ELISA analysis in association with other endpoints.
Chronic changes in concentration of plasma and serum biomarkers | 4 weeks
  Biomarkers of insulin, glucose, cholesterol and resveratrol metabolites will be measured in plasma and serum using liquid chromatography-mass spectrometry and ELISA analysis in association with other endpoints.
Acute and chronic changes in blood pressure | 1 hour post dose, 4 weeks
  Systolic and diastolic blood pressure will be taken after each cognitive assessment (measured in mm Hg).
Acute and chronic changes in heart rate | 1 hour post dose, 4 weeks
  Heart rate will be measured after each cognitive assessment (measured in BPM).
Changes in weight and Body Mass Index (BMI) | 4 weeks
  Participants weight will be recorded at testing visits and BMI will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Wightman, Dr, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom